### Is it really necessary going all over the top in patients with symptomatic lumbar canal stenosis?

Non-inferiority of osseous decompression of the lumbar canal until normalization of epidural pressure compared to conventional open laminectomy in patients with symptomatic lumbar canal stenosis.

24/605-EC-X Tesis

June 2, 2025

Juan Pablo Castaño Montoya
Universidad Complutense de Madrid
+34-669345474
juanpablo.castano@salud.madrid.org

### 1. Terminology

- Pressure-guided laminectomy (PGL): Bone resection of the lamina and ligamentum flavum until epidural pressure reaches a normal value in the stenotic segment.
- Non-pressure-guided laminectomy (NPGL): Complete resection of both the lamina and ligamentum flavum in the stenotic segment.

### 2. Introduction

Lumbar spinal canal stenosis is a prevalent and disabling cause of low back and lower limb pain in the elderly, and it is estimated to affect over 103 million people worldwide. (1) It significantly impairs patients' quality of life due to the presence of pain and gait disturbances, impacting social functioning and contributing to the development of psychological disorders. (2) Three main hypotheses have been proposed to explain the phenomenon of neurogenic claudication: the postural theory, the ischemic theory, and the venous stasis theory. However, the precise mechanism by which nerve root compression causes the typical clinical presentation of lumbar stenosis remains incompletely understood. (3)

A wide range of therapeutic options exists for the management of lumbar spinal stenosis, from conservative treatments such as physical therapy and neuromodulators to percutaneous procedures like epidural injections, and finally surgical approaches ranging from decompression to spinal fusion (1,4). Current surgical techniques focus on decompressing the dural sac to address a mechanical compression problem. These procedures can be performed through open surgery or minimally invasive methods using endoscopic or tubular approaches.

A study conducted at this hospital by Carrascosa et al., with results published in 2020 and 2023, found that in patients who underwent canal decompression via laminectomy with radiologic confirmation of the dural sac decompression area, clinical improvement was not associated with the postoperative area of the spinal canal or thecal sac (5,6). Similar findings have been reported in other studies, emphasizing the poor clinicoradiological correlation in this condition, which suggests that the pathogenesis of lumbar spinal stenosis may not be solely mechanical, and that additional contributing factors may be involved (7–9).

Our research group has developed an interest in identifying these additional factors and has proposed a new theory to explain neurogenic claudication. We hypothesize that epidural pressure is elevated in stenotic segments compared to healthy ones and plays a role in the disease's pathophysiology, either by impairing cerebrospinal fluid (CSF) flow or by causing local ischemia of the cauda equina nerve roots. This is supported by evidence of increased epidural pressure

in patients with spinal stenosis compared to healthy controls, as well as the observation of dynamic epidural pressure changes in patients with neurogenic claudication (10–12).

This theory supports the use of minimally invasive procedures, which aim to decompress the canal through small access corridors without requiring open surgery, extensive dissection of the lumbar musculature, or resection of bone and ligamentous structures. In this way, it is possible to minimize the risk of secondary spinal instability by performing decompression through a unilateral approach while preserving midline structures such as the supraspinous and interspinous ligaments and the paravertebral musculature (13–16).

Based on the aforementioned rationale, this study aims to evaluate the non-inferiority of pressure-guided lumbar canal decompression—until epidural pressure normalizes in the stenotic segment—compared to conventional open laminectomy without pressure guidance. Both groups will be assessed using clinical scales and radiologic imaging to determine clinical improvement. We hope that the results of this study will support the theory of lumbar epidural hypertension as a potential etiological factor in neurogenic claudication.

### 3. Hypothesis

The null hypothesis is that non-inferiority of pressure-guided laminectomy compared to non-pressure-guided laminectomy cannot be demonstrated in patients diagnosed with symptomatic lumbar spinal stenosis.

The alternative hypothesis is that osseous decompression of the lumbar canal until epidural pressure normalization is not inferior to conventional open laminectomy in achieving clinical improvement in patients with symptomatic lumbar spinal stenosis, as measured by the Zurich Claudication Questionnaire (ZCQ).

### 4. Objectives

### 4.1. General objective

To assess whether osseous decompression of the lumbar canal until normalization of epidural pressure is not inferior to conventional open laminectomy in achieving clinical improvement in patients with symptomatic lumbar spinal stenosis, as measured by the clinical severity subscale of the Zurich Claudication Questionnaire (ZCQ).

### 4.2. Specific objetives

- To characterize the demographic variables of patients undergoing surgical treatment for lumbar spinal stenosis.
- To compare the clinical response of patients treated using the two different surgical techniques.
- To determine the extent of osseous decompression performed using imaging techniques.
- To evaluate the complications associated with the surgical procedures.

#### 5. Materials and methods

A single-blind, randomized, controlled non-inferiority clinical trial is proposed to compare the effectiveness of total osseous decompression of the lumbar canal until normalization of epidural pressure versus conventional open laminectomy in patients with symptomatic lumbar spinal stenosis.

### 5.1. Study and reference population

The study will include patients with chronic low back pain and/or lower limb pain secondary to lumbar spinal canal stenosis, who are treated at the San Carlos Clinical Hospital and attend consultations in the Neurosurgery Department. Given the vulnerability of the study population, an a priori sample size calculation will be performed to ensure the objectives can be met and a representative sample of this patient population can be obtained.

To improve the statistical reliability of the study results, a minimum sample of 24 subjects has initially been selected. The study will be conducted in the Neurosurgery Department at the San Carlos Clinical Hospital in Madrid.

### 5.2. Inclusion and exclusion criteria

Inclusion criteria:

- Age over 50 years.
- Surgical indication determined by:
  - Low back and/or lower limb pain lasting more than 3 months.
  - Pain refractory to conservative medical treatment (analgesics, physical therapy, epidural block).
  - Clinical criterion for neurogenic claudication defined as a score ≥11 on the N-CLASS scale (Annex 1). (17)
  - o Preoperative MRI confirming spinal canal stenosis. (18)
- Patient agrees to undergo the proposed surgical intervention.
- Patient consents to participate in the study by signing the informed consent form.

#### Exclusion criteria:

- Foraminal or lateral recess stenosis.
- Symptomatic disc herniation at the surgical level.
- Spondylolisthesis greater than Meyerding Grade I (vertebral displacement >25%) or spondylolysis.
- Radiological instability defined as sagittal plane displacement >5 mm on dynamic flexion-extension spinal X-rays.
- Scoliosis with a Cobb angle >30°.
- Compression fracture at the target surgical level.
- Previous surgery at the same level to be treated.
- Prior infection at the target level.
- Contraindication for magnetic resonance imaging.
- Diagnosis of major depression or dysthymia according to DSM-V criteria.
   (19)

### 5.3. Withdrawal criteria

- The patient requests to withdraw from the study.
- Inability to follow the assigned surgical protocol (e.g., intraoperative necessity to convert to a different surgical technique due to unforeseen findings).
- Medical events that contraindicate surgical intervention.
- Withdrawal of informed consent by the patient.

### 5.4. Dropouts and management of withdrawals

Patients who choose to withdraw from the study may do so at any time without any negative consequences to their medical care.

Data collected up to the point of withdrawal will be used for analytical purposes unless the patient explicitly requests otherwise. Confidentiality and current data protection regulations will be always respected.

### 5.5. Study Termination

The study will conclude once follow-up of all enrolled patients has been completed and the required sample size for statistical analysis has been achieved.

Likewise, the study may be terminated early by decision of the ethics committee or the principal investigators if unforeseen risks are identified or if insurmountable difficulties in conducting the study arise.

### 5.6. Sample size

The sample size was estimated using the TwoSampleMean.NIS function from the **TrialSize** package of the statistical software R v.4.4.0. The expected mean difference between the groups in the ZCQ clinical severity subscale is 0.51 with a standard deviation of 0.57. With a non-inferiority margin set at 0.75 (minimal clinically important difference), a one-sided  $\alpha$  of 0.05, and a  $\beta$  of 0.20, we estimate that a sample size of 20 patients would demonstrate non-inferiority with a power of 80%. Finally, based also on similar previous studies and considering a dropout rate of 20%, we decided to assume a total N of 24 patients to justify a sample size capable of meeting the general study objectives. (20,21)

### 6. Experimental design

### 6.1. Study design and work plan

A single-blind, randomized, controlled non-inferiority clinical trial will be conducted to compare the effectiveness of total osseous decompression of the lumbar canal until normalization of epidural pressure versus open laminectomy in patients with symptomatic lumbar spinal stenosis.

The study will not involve participation from the medical industry, and the research protocol will be registered on ClinicalTrials.gov.

The indication for surgical intervention will be made by a single neurosurgeon from the San Carlos Clinical Hospital, based on clinical scales and imaging studies as outlined in the inclusion criteria. After signing the informed consent form (Annex 2) and being included on the surgical waiting list, patients will be randomized 1:1 using a simple randomization method implemented through SPSS software. Baseline evaluations will include various clinical scales (ZCQ, Numeric Pain Rating Scale [NPRS], Oswestry Disability Index [ODI], and Japanese Orthopedic Association Back Pain Evaluation Questionnaire [JOABPEQ]). The patient will remain blinded to their assigned surgical intervention.

### Study interventions (Figure 1):

• Non-Pressure-Guided Laminectomy (NPGL): Open laminectomy with total decompression of the posterior elements. This is defined as the classical technique, in which, after muscle dissection, a Codman microsensor (Integra LifeSciences) will be inserted into the epidural space under direct visualization. Careful dissection of the ligamentum flavum below the right hemilamina will be performed to obtain the patient's baseline epidural pressure (Figure 2). The sensor will then

be removed, and resection of the spinous process, supraspinous and interspinous ligaments, hemilaminae, and ligamentum flavum will be carried out bilaterally until proper decompression of the thecal sac is visualized.

# • Pressure-Guided Laminectomy (PGL): After muscle dissection, the Codman microsensor will be inserted into the lower epidural space as described above. The patient's baseline epidural pressure will be recorded, and osseous decompression will begin following the "unilateral laminotomy for bilateral decompression" technique from the left side, continuing until epidural pressure decreases to 10 mmHg—previously established as a median non-pathological value

(22,23).



Figura 1. Schematic of the osseous decompression to be performed during surgical interventions (adapted figure). (24)



Figura 2. A. Codman Microsensor. B. Codman ICP Express Monitor. C. Technique for inserting the pressure catheter into the epidural space at the stenotic level.

The CODMAN MICROSENSOR pressure catheter (Integra LifeSciences) is a transducer with a micro-strain gauge at its distal end that records pressure changes in a medium. At the proximal end, it has an electrical connector that must be linked to the ICP-EXPRESS monitor. This sensor model was chosen due to its availability in the operating room and its prior use in published scientific studies. (11)

All procedures will be performed by a single neurosurgeon from the San Carlos Clinical Hospital. Patients will be evaluated two weeks postoperatively, during which clinical scales will be applied, and the surgical wound will be assessed. Follow-up will continue at 3 and 6 months via telephone, and at 12 months in person to reassess clinical outcomes.

Additionally, a follow-up lumbar MRI will be performed 3 months after surgery to evaluate the degree of decompression achieved.

### 6.2. Data collection and information sources

Sociodemographic data and clinical outcome variables will be collected during the preoperative consultation and during follow-up visits at 1, 3, and 6 months, as well as at one-year post-surgery. Imaging data will be obtained from the patient's preoperative (baseline) lumbar spine MRI and from a follow-up MRI performed three months after the surgical procedure. T2-weighted axial sequences will be used to assess the degree of osseous decompression achieved.

### 6.3. Variables

### 6.3.1. Outcome variables

- Primary outcome: ZCQ Symptom Severity Subscale (Annex 4): consists
  of 7 items assessing symptom severity over the past month using a 5-point
  numerical scale, where 5 indicates greater severity. The final score is
  calculated as the mean of all item scores. (28–33)
- Secondary outcomes:
  - ZCQ Physical Function Subscale (Annex 4): consists of 5 items evaluating functional impairment over the past month on a 4-point scale, where 4 indicates greater disability. The mean score of the items is used as the result. (28,31,33–35)
  - ZCQ Patient Satisfaction Subscale (Annex 4): consists of 5 items categorized into 4 levels (from very satisfied to very dissatisfied). It evaluates overall outcome, pain relief, walking capacity, ability to work, perform household or gardening tasks, strength, and balance. This subscale will be applied at 6 and 12 months postoperatively. (28,31,33)
  - NPRS (Annex 5): The Numeric Pain Rating Scale is an 11-point scale in which patients rate their pain from 0 to 10, with 0 (on the left) representing "no pain" and 10 (on the right) representing "worst imaginable pain." It will assess both lower limb symptoms (NPRS lower limbs) and low back and/or gluteal pain (NPRS back or gluteal region). (36,37)
  - ODI (Annex 6): The Oswestry Disability Index assesses pain-related disability across 10 items; each scored from 0 (normal) to 5 (severely affected). The final score is calculated as the sum of item scores divided by the total possible score and multiplied by 100. Disability is classified as: mild (0–20%), moderate (21–40%), severe (41–60%), crippled (61–80%), and bed-bound or symptom exaggeration (>80%). (30,38–40)
  - JOABPEQ (Annex 7): The Japanese Orthopedic Association Back Pain Evaluation Questionnaire includes five domains: pain-related disorders, lumbar dysfunction, gait disturbance, impairment of

social life, and psychological disorders. Scores range from 0 to 100, with higher scores indicating better health status. (2,41)

- Surgical complications.
- o Reoperation.

### 6.3.2. Variables of interest

- Sociodemographic:
  - o Age.
  - o Gender.
  - Marital status.
  - Social risk factor (defined as poor family support or undergoing disability benefit procedures)

### Clinical:

- o Duration of symptoms (in months).
- o Pain location (lumbar, lower limbs, or both).
- o Predominant pain type (axial or appendicular).
- Smoking history.
- o Overweight (BMI > 25).
- Opioid dosage (expressed in morphine milligram equivalents). (25)

### Imagen:

- Preoperative MRI:
  - Degree of lumbar canal stenosis according to the Schizas morphological classification (Annex 3). (26)
- Postoperative MRI:
  - Degree of decompression based on the dural sac crosssectional area (DSCA) (Figure 3) (24,27)



Figure 3. Measurement of the dural sac cross-sectional area before (left) and after decompressive surgery (right) in patients with lumbar spinal stenosis. (9)

### 6.4. Data management

The database generated by the study will not contain any patient-identifying information; patient identity will remain confidential. Study data will be recorded in a dissociated manner and linked to a code assigned to each patient, so that only the investigator can associate the data with a clinical record. Only the investigators and personnel responsible for ensuring data quality and analysis will have access to participants' clinical documentation.

The study will comply with Regulation (EU) 2016/679 of the European Parliament and of the Council of 27 April 2016, concerning the protection of natural persons with regard to the processing of personal data and the free movement of such data, and repealing Directive 95/46/EC (General Data Protection Regulation), as well as with the Spanish Organic Law 3/2018 of 5 December on the Protection of Personal Data and the Guarantee of Digital Rights (LOPDGDD).

The data controller is the San Carlos Clinical Hospital. Its data protection officer is the DPO Committee of the Health Department of the Community of Madrid, which will process the data for the purposes indicated in this document.

Personal data, including health information, will be retained for the duration of the project and for up to three years after its conclusion. Patients may exercise their rights to access and rectify their data, as well as their right to restrict data processing and to request a copy of the data or to have it transferred to a third party.

### 6.5. Study populations

- 6.5.1. Per protocol population (PP): Includes all patients who completed all scheduled visits and strictly adhered to the study protocol instructions.
- 6.5.2. Intention-to-treat population (ITT): Includes all patients who were initially assigned to an intervention group, regardless of whether they deviated from the protocol.

### 6.6. Data analysis

The demographic and clinical data of the study will be described using descriptive statistical indices. Quantitative variables will be summarized using the mean and standard deviation (SD). For quantitative variables that do not follow a normal

distribution, the median and interquartile range (IQR) will be reported. Qualitative variables will be presented as frequency distributions.

No interim efficacy analysis will be conducted.

The efficacy analysis will be performed using both the Per-Protocol (PP) and Intention-To-Treat (ITT) populations. The safety analysis will be performed exclusively on the ITT population. Data will be analyzed longitudinally, and the primary analysis will focus on differences in effectiveness, measured using the ZCQ scale and other clinical outcome measures, between the two surgical intervention groups. Interactions between treatment and time will also be examined to explore potential temporal variations in the treatment effect.

Non-inferiority analysis will be carried out using linear regression models, applying a one-sided significance level ( $\alpha$ ) of 0.05 and the non-inferiority margins detailed in Table 1. (20,21,42–46). Multiple non-inferiority hypotheses (one for each clinical scale) will be evaluated. Statistical adjustment for multiplicity will be applied to control the overall type I error rate, progressively narrowing the allowable error margin to maintain the required global error threshold across all comparisons.

**Table 1. Non-inferiority margins.** 

| Outcome | Expected difference | Non-inferiority margin |
|-------------------------|---------------------|------------------------|
| ZCQ (symptom severity) | 0,7 | 0,75 |
| ZCQ (physical function) | 0,6 | 0,6 |
| NRPS back or gluteal | 2 | 1,25 |
| NRPS lower extremity | 2 | 1,5 |
| ODI | 10 | 5 |
| JOABPEQ | 20 | 20 |

In addition to unadjusted models, all analyses will also be adjusted for potential confounding variables such as age, sex, and comorbidities using multiple linear regression.

The safety analysis will examine the complications that occur during the study period. Their association with the surgical intervention will be analyzed using logistic regression models. For these analyses, a two-sided significance level ( $\alpha$ ) of 0.05 will be used.

All results will be presented as point estimates with corresponding 95% confidence intervals (CIs). These estimates will be compared against the predefined non-inferiority margins to determine whether non-inferiority can be established. All statistical analyses will be performed using IBM SPSS Statistics version 26 and R version 4.4.1.

### 6.7. Resources

- Human resources:
  - Neurosurgeon.
  - Neurosurgery Resident Physician.
  - UAMI (Unit for Methodological Support in Research).
- Facilities:
  - Scheduled surgery operating room.
  - Outpatient consultation room equipped with a chair, desk, computer, and examination table.
  - Office with a computer workstation.
- Specialized Equipment:
  - o Intracranial pressure monitoring catheter (Codman).
  - o Intracranial pressure monitoring device.

### 6.8. Timeline

The estimated duration of the trial is two years, subdivided into a 12-month patient recruitment period and one year of follow-up.



### 6.9. Adverse events

It is the responsibility of the investigator to detect and document any event that meets the criteria and definitions of an adverse event (AE). All AEs will be reported in accordance with the guidelines set forth in the "CONSORT Statement for Randomized Trials of Nonpharmacologic Treatments: A 2017 Update and a CONSORT Extension for Nonpharmacologic Trial Abstracts."" (47)

#### 6.10. Ethical considerations

The clinical trial will be conducted in accordance with the principles outlined in the Declaration of Helsinki (Annex IV), as well as the current legal regulations in force in Spain. The study will commence only after obtaining approval from the relevant Clinical Research Ethics Committee (CEIC).

### 6.11. Dissemination plan

Once the study is completed, the results will be prepared for publication in national or international scientific journals and for presentation at conferences. The principal investigator commits to complying with current Spanish legislation, which mandates the publication of results—whether positive or negative—in scientific journals. The publications will acknowledge the Clinical Research Ethics Committee (CEIC) that approved the study and disclose the source of funding.

### 7. References

- 1. Katz JN, Zimmerman ZE, Mass H, Makhni MC. Diagnosis and Management of Lumbar Spinal Stenosis: A Review. JAMA. 3 de mayo de 2022;327(17):1688-99.
- 2. Kobayashi H, Sekiguchi M, Yonemoto K, Kakuma T, Tominaga R, Kato K, et al. Reference values of the Japanese Orthopaedic Association Back Pain Evaluation Questionnaire in patients with lumbar spinal stenosis and characteristics of deterioration of QOL: Lumbar Spinal Stenosis Diagnosis Support Tool: DISTO project. J Orthop Sci. julio de 2019;24(4):584-9.
- 3. Chad DA. Lumbar spinal stenosis. Neurol Clin. mayo de 2007;25(2):407-18.
- 4. Chen X, Zheng Z, Lin J. Clinical Effectiveness of Conservative Treatments on Lumbar Spinal Stenosis: A Network Meta-Analysis. Front Pharmacol. 2022;13:859296.
- 5. Carrascosa-Granada A, Velazquez W, Wagner R, Saab Mazzei A, Vargas-Jimenez A, Jorquera M, et al. Comparative Study Between Uniportal Full-Endoscopic Interlaminar and Tubular Approach in the Treatment of Lumbar Spinal Stenosis: A Pilot Study. Global Spine J. abril de 2020;10(2 Suppl):70S-78S.
- 6. Süner HI, Castaño JP, Vargas-Jimenez A, Wagner R, Mazzei AS, Velazquez W, et al. Comparison of the Tubular Approach and Uniportal Interlaminar Full-Endoscopic Approach in the Treatment of Lumbar Spinal Stenosis: Our 3-Year Results. World Neurosurgery. 1 de mayo de 2023;173:e148-55.
- 7. Boden SD, Davis DO, Dina TS, Patronas NJ, Wiesel SW. Abnormal magnetic-resonance scans of the lumbar spine in asymptomatic subjects. A prospective investigation. J Bone Joint Surg Am. marzo de 1990;72(3):403-8.
- 8. Gupta S, Bansal T, Kashyap A, Sural S. Correlation between clinical scoring systems and quantitative MRI parameters in degenerative lumbar spinal stenosis. J Clin Orthop Trauma. diciembre de 2022;35:102050.
- 9. Hermansen E, Myklebust TÅ, Weber C, Brisby H, Austevoll IM, Hellum C, et al. Postoperative Dural Sac Cross-Sectional Area as an Association for Outcome After Surgery for Lumbar Spinal Stenosis: Clinical and Radiological Results From the NORDSTEN-Spinal Stenosis Trial. Spine (Phila Pa 1976). 15 de mayo de 2023;48(10):688-94.
- 10. Takahashi K, Kagechika K, Takino T, Matsui T, Miyazaki T, Shima I. Changes in epidural pressure during walking in patients with lumbar spinal stenosis. Spine (Phila Pa 1976). 15 de diciembre de 1995;20(24):2746-9.
- 11. Barz T, Melloh M, Staub LP, Lord SJ, Lange J, Merk HR. Increased intraoperative epidural pressure in lumbar spinal stenosis patients with a positive nerve

- root sedimentation sign. Eur Spine J. mayo de 2014;23(5):985-90.
- 12. Takahashi K, Miyazaki T, Takino T, Matsui T, Tomita K. Epidural pressure measurements. Relationship between epidural pressure and posture in patients with lumbar spinal stenosis. Spine (Phila Pa 1976). 15 de marzo de 1995;20(6):650-3.
- 13. Boukebir MA, Berlin CD, Navarro-Ramirez R, Heiland T, Schöller K, Rawanduzy C, et al. Ten-Step Minimally Invasive Spine Lumbar Decompression and Dural Repair Through Tubular Retractors. Oper Neurosurg (Hagerstown). 1 de abril de 2017;13(2):232-45.
- 14. Soliman MAR, Ali A. Decompression of lumbar canal stenosis with a bilateral interlaminar versus classic laminectomy technique: a prospective randomized study. Neurosurg Focus. 1 de mayo de 2019;46(5):E3.
- 15. Zhang C, Chen L, Li J, Huang D, Zhang W, Lin J. Should Posterior Midline Structures Be Preserved in Decompression Surgery for Lumbar Spinal Stenosis?: A Systematic Review and Meta-analysis. Clin Spine Surg. 1 de octubre de 2022;35(8):341-9.
- 16. Mariconda M, Fava R, Gatto A, Longo C, Milano C. Unilateral laminectomy for bilateral decompression of lumbar spinal stenosis: a prospective comparative study with conservatively treated patients. J Spinal Disord Tech. febrero de 2002;15(1):39-46.
- 17. Genevay S, Courvoisier DS, Konstantinou K, Kovacs FM, Marty M, Rainville J, et al. Clinical classification criteria for neurogenic claudication caused by lumbar spinal stenosis. The N-CLASS criteria. Spine J. junio de 2018;18(6):941-7.
- 18. Steurer J, Roner S, Gnannt R, Hodler J. Quantitative radiologic criteria for the diagnosis of lumbar spinal stenosis: a systematic literature review. BMC Musculoskelet Disord. 28 de julio de 2011;12:175.
- 19. American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders [Internet]. 5th ed. Washington, DC; 2013. Disponible en: http://dx.doi.org/10.1176/appi.books.9780890425596
- 20. Cleland JA, Whitman JM, Houser JL, Wainner RS, Childs JD. Psychometric properties of selected tests in patients with lumbar spinal stenosis. Spine J. octubre de 2012;12(10):921-31.
- 21. Fukushima M, Oka H, Oshima Y, Yuzawa Y, Matsudaira K, Tanaka S, et al. Evaluation of the Minimum Clinically Important Differences of the Zurich Claudication Questionnaire in Patients With Lumbar Spinal Stenosis. Clin Spine Surg. diciembre de 2020;33(10):E499-503.
- 22. Spetzger U, Bertalanffy H, Naujokat C, von Keyserlingk DG, Gilsbach JM. Unilateral laminotomy for bilateral decompression of lumbar spinal stenosis. Part I: Anatomical and surgical considerations. Acta Neurochir (Wien). 1997;139(5):392-6.
- 23. Jia R, Wang XQ, Zhang Y, Hsueh S. Long-Term Outcomes After Minimally Invasive Bilateral or Unilateral Laminotomy for Degenerative Lumbar Spinal Stenosis: A Minimum 10-Year Follow-Up Study. World Neurosurg. agosto de 2022;164:e1001-6.
- 24. Hermansen E, Austevoll IM, Hellum C, Storheim K, Myklebust TÅ, Aaen J, et al. Comparable increases in dural sac area after three different posterior decompression techniques for lumbar spinal stenosis: radiological results from a randomized controlled trial in the NORDSTEN study. Eur Spine J. septiembre de 2020;29(9):2254-61.
- 25. Dowell D, Haegerich TM, Chou R. CDC Guideline for Prescribing Opioids for Chronic Pain--United States, 2016. JAMA. 19 de abril de 2016;315(15):1624-45.
- 26. Schizas C, Theumann N, Burn A, Tansey R, Wardlaw D, Smith FW, et al. Qualitative grading of severity of lumbar spinal stenosis based on the morphology of the dural sac on magnetic resonance images. Spine (Phila Pa 1976). 1 de octubre de

- 2010;35(21):1919-24.
- 27. Hermansen E, Myklebust TÅ, Austevoll IM, Hellum C, Storheim K, Banitalebi H, et al. Dural Sac Cross-sectional area change from preoperatively and up to 2 years after decompressive surgery for central lumbar spinal stenosis: investigation of operated levels, data from the NORDSTEN study. Eur Spine J. 8 de abril de 2024;
- 28. Stucki G, Daltroy L, Liang MH, Lipson SJ, Fossel AH, Katz JN. Measurement Properties of a Self-Administered Outcome Measure in Lumbar Spinal Stenosis. Spine [Internet]. 1996;21(7). Disponible en:
- https://journals.lww.com/spinejournal/fulltext/1996/04010/measurement\_properties\_of\_a\_self\_administered.4.aspx
- 29. Comer CM, Conaghan PG, Tennant A. Internal construct validity of the Swiss Spinal Stenosis questionnaire: Rasch analysis of a disease-specific outcome measure for lumbar spinal stenosis. Spine (Phila Pa 1976). 1 de noviembre de 2011;36(23):1969-76.
- 30. Tonosu J, Takeshita K, Hara N, Matsudaira K, Kato S, Masuda K, et al. The normative score and the cut-off value of the Oswestry Disability Index (ODI). Eur Spine J. agosto de 2012;21(8):1596-602.
- 31. Hidalgo Ovejero AM, Menéndez García M, Bermejo Fraile B, García Mata S, Forcén Alonso T, Mateo Sebastián P. Cross-cultural adaptation of the Zurich Claudication Questionnaire. Validation study of the Spanish version. An Sist Sanit Navar. abril de 2015;38(1):41-52.
- 32. Fujimori T, Ikegami D, Sugiura T, Sakaura H. Responsiveness of the Zurich Claudication Questionnaire, the Oswestry Disability Index, the Japanese Orthopaedic Association Back Pain Evaluation Questionnaire, the 8-Item Short Form Health Survey, and the Euroqol 5 dimensions 5 level in the assessment of patients with lumbar spinal stenosis. Eur Spine J. junio de 2022;31(6):1399-412.
- 33. Wertli MM, Rossi D, Burgstaller JM, Held U, Ulrich NH, Farshad M, et al. Validity of outcome measures used in randomized clinical trials and observational studies in degenerative lumbar spinal stenosis. Sci Rep. 19 de enero de 2023;13(1):1068.
- 34. Tomkins CC, Battié MC, Hu R. Construct validity of the physical function scale of the Swiss Spinal Stenosis Questionnaire for the measurement of walking capacity. Spine (Phila Pa 1976). 1 de agosto de 2007;32(17):1896-901.
- 35. Araki M, Nonoshita H, Kitano S, Shigematsu H, Tanaka M, Kawasaki S, et al. The critical cutoff point of the Zurich Claudication Questionnaire and the Japanese Orthopaedic Association score indicating locomotive syndrome in patients with lumbar spinal canal stenosis. J Orthop Sci. marzo de 2021;26(2):290-4.
- 36. Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine (Phila Pa 1976). 1 de junio de 2005;30(11):1331-4.
- 37. Chiarotto A, Maxwell LJ, Ostelo RW, Boers M, Tugwell P, Terwee CB. Measurement Properties of Visual Analogue Scale, Numeric Rating Scale, and Pain Severity Subscale of the Brief Pain Inventory in Patients With Low Back Pain: A Systematic Review. J Pain. marzo de 2019;20(3):245-63.
- 38. Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 15 de noviembre de 2000;25(22):2940-52; discussion 2952.
- 39. Pratt RK, Fairbank JCT, Virr A. The reliability of the Shuttle Walking Test, the Swiss Spinal Stenosis Questionnaire, the Oxford Spinal Stenosis Score, and the Oswestry Disability Index in the assessment of patients with lumbar spinal stenosis. Spine (Phila Pa 1976). 1 de enero de 2002;27(1):84-91.
- 40. Vishwanathan K, Braithwaite I. Construct validity and responsiveness of commonly used patient reported outcome instruments in decompression for lumbar

- spinal stenosis. J Clin Orthop Trauma. mayo de 2021;16:125-31.
- 41. Fukui M, Chiba K, Kawakami M, Kikuchi S ichi, Konno S ichi, Miyamoto M, et al. Japanese Orthopaedic Association Back Pain Evaluation Questionnaire. Part 3. Validity study and establishment of the measurement scale: Subcommittee on Low Back Pain and Cervical Myelopathy Evaluation of the Clinical Outcome Committee of the Japanese Orthopaedic Association, Japan. J Orthop Sci. mayo de 2008;13(3):173-9.
- 42. Ostelo RWJG, Deyo RA, Stratford P, Waddell G, Croft P, Von Korff M, et al. Interpreting change scores for pain and functional status in low back pain: towards international consensus regarding minimal important change. Spine (Phila Pa 1976). 1 de enero de 2008;33(1):90-4.
- 43. Haase I, Kladny B. Clinical Relevance of Changes in Pain Intensity in Patients with Specific Back Pain. Z Orthop Unfall. abril de 2022;160(2):213-21.
- 44. Ogura Y, Ogura K, Kobayashi Y, Kitagawa T, Yonezawa Y, Takahashi Y, et al. Minimally clinically important differences for the Japanese Orthopaedic Association Back Pain Evaluation Questionnaire (JOABPEQ) following decompression surgery for lumbar spinal stenosis. J Clin Neurosci. noviembre de 2019;69:93-6.
- 45. Fujimori T, Miwa T, Oda T. Responsiveness of the Japanese Orthopaedic Association Back Pain Evaluation Questionnaire in lumbar surgery and its threshold for indicating clinically important differences. Spine J. enero de 2019;19(1):95-103.
- 46. Takenaka H, Kamiya M, Sugiura H, Nishihama K, Suzuki J, Hanamura S. Recovery of the Japanese orthopedic association back pain evaluation questionnaire score and walking ability following lumbar spinal stenosis surgery. Eur Spine J. 7 de abril de 2024;
- 47. Boutron I, Altman DG, Moher D, Schulz KF, Ravaud P. CONSORT Statement for Randomized Trials of Nonpharmacologic Treatments: A 2017 Update and a CONSORT Extension for Nonpharmacologic Trial Abstracts. Ann Intern Med. 4 de julio de 2017;167(1):40-7.

### Annex 1. N-CLASS criteria.

Neurogenic claudication caused by lumbar spinal stenosis score (simplified weighted score)

| Age >60 y | 4 |
|-----------------------------------------------|---|
| Positive 30-s extension test | 4 |
| Patient reports pain in both legs | 3 |
| Patient reports leg pain relieved by sitting | 3 |
| Patient reports leg pain decreased by leaning | 3 |
| forward or flexing the spine | |
| Negative SLR-60 test | 2 |

SLR-60, straight leg raise test is positive if leg pain is produced below  $60^{\circ}$ .

### Annex 2. Informed consent.

### INFORMED CONSENT FOR LAMINECTOMY AND EPIDURAL PRESSURE RECORDING

### **PARTICIPATION IN THE STUDY**

You are invited to participate in the study titled: "Non-inferiority of osseous decompression of the lumbar canal until normalization of epidural pressure compared to conventional open laminectomy in patients with symptomatic lumbar canal stenosis." You have the right to be informed about the procedures to which you will be subjected and the potential complications that may arise. This document aims to explain all these issues. Please read it carefully and consult your Neurosurgeon with any questions that may arise.

We remind you that, for legal reasons, you or your legal representative, if applicable (family member or person with close personal ties), must sign the Informed Consent in order for the surgical procedure to be carried out.

It is important to understand that participation in this study is voluntary. Once you give your consent to be included in the study, you may withdraw it at any time without this affecting your medical care.

Lumbar canal stenosis is a prevalent and disabling cause of lower back and leg pain and is associated with a significant decline in patients' quality of life due to pain and gait impairment. It is defined as narrowing of the spinal canal in the lumbar area, which compresses the spinal nerves traveling to the legs. The diagnosis is established by the presence of characteristic symptoms and confirmed through imaging studies (MRI).

Although multiple theories attempt to explain the effects caused by this disease, the exact mechanism remains unknown. Through this study, our group aims to evaluate the epidural pressure theory by comparing a surgical intervention involving less bone removal to the conventional surgery, with the goal of preventing future mechanical instability of the lumbar spine.

Both surgical procedures are performed under general anesthesia. Access to the affected level will be via a posterior approach to the spine. The procedure involves bone resection at the back of the vertebra to remove excess bone and ligaments and ensure decompression of the dural sac, the structure that covers the lumbar nerves.

By agreeing to participate in the study, you consent to the use of personal clinical and radiological data for analysis, always maintaining the confidentiality of personal data (Annex: confidentiality and data protection).

#### **DESCRIPTION OF STUDY PROCEDURES**

By agreeing to participate in this study, you acknowledge that you will be randomized to receive one of the following procedures:

- Open Laminectomy: This consists of the removal of the bony structures of the vertebrae known as spinous processes and laminae, along with the supraspinous and interspinous ligaments and the ligamentum flavum located between the laminae and the membrane covering the nerve roots (dura mater), to decompress the neural structures.
- Unilateral Laminotomy for Bilateral Open Decompression: This involves the
  resection of the vertebral laminae and ligamentum flavum located between them
  and the dura mater, with the aim of decompressing the neural structures. The
  bone resection will be performed from one side only, intending to remove the
  necessary bone to normalize the pressure on the neural structures. The following
  structures will be preserved: spinous process, supraspinous and interspinous
  ligaments, to minimize postoperative segmental instability.

Additionally, the study includes the measurement of epidural pressure at the affected level causing symptoms, before performing the laminectomy and both before and during the laminotomy. This will be done by inserting a pressure microsensor between the ligamentum flavum and the dura mater once the vertebral level has been identified during surgery. The sensor will be removed after pressure measurement in the laminectomy and after completing bone decompression in the laminotomy. These steps do not carry significant surgical risk. During the study, you will not know whether bone resection was guided by pressure measurement and may find out once follow-up is complete or if you choose to withdraw from the study.

### **PREOPERATIVE**

Before surgery, you will need to undergo blood tests, a chest X-ray, and an ECG. You will also have a pre-anesthesia assessment and receive preoperative instructions (fasting hours, medication adjustments, etc.).

### POSSIBLE RISKS, DISCOMFORTS, AND CONSEQUENCES

After surgery, you may experience pain at the incision site that may last several weeks. You should know that lumbar stenosis is a degenerative spinal process strongly associated with aging, and that surgery will decompress the lumbar nerves but will not restore the spine to its prior condition. Pain relief is expected, but complete resolution is not guaranteed.

After recovering from anesthesia, the patient will be admitted to the general neurosurgery ward or intensive care unit if required. You will then gradually resume walking with assistance. If there are no complications, discharge will occur within 1 to 3 days. You will return after two weeks for wound care follow-up and suture removal if appropriate.

### **POSSIBLE COMPLICATIONS**

You should know that every surgical procedure carries potential complications due to the technique itself and individual factors (diabetes, heart disease, hypertension, anemia, obesity, etc.). These may require additional medical or surgical treatment and, in rare cases, can result in death.

### Main complications include:

- 1. Spinal cord or nerve root injury: May cause paralysis, sensory deficits, or loss of bladder/bowel control, which may be temporary or permanent.
- 2. Dura mater injury or rupture: Can occur during surgery or epidural pressure catheter insertion. Even with intraoperative repair, a cerebrospinal fluid leak may develop, requiring bed rest for 5 days or a new surgical procedure.
- 3. Venous thrombosis in the lower limbs: May lead to leg swelling and, rarely, pulmonary embolism, which can be fatal.
- 4. Bleeding: May be superficial or deep and occasionally require surgical evacuation.
- 5. Surgical wound infection: May be superficial or deep and may require reoperation. Can also lead to cerebrospinal fluid infection (meningitis), requiring long-term antibiotics.

#### **ALTERNATIVE TREATMENTS**

Alternatives include conventional open laminectomy or continuation of medical treatment: analgesics, anti-inflammatories, lumbosacral orthosis, epidural injections, and rehabilitation.

#### **BENEFITS**

It is possible that none of the surgical interventions will improve symptoms. When improvement occurs, it usually lasts up to 4 years post-surgery. The new surgical technique aims to achieve similar clinical improvement with less bone resection, potentially reducing future spinal instability. Your participation will also provide data that may benefit other patients in the future.

### PATIENT'S DECLARATION

After receiving this information, the patient or legal representative **HEREBY DECLARES**:

- 1. Having received clear and precise information from the physician about the personalized risks and alternatives.
- 2. Being satisfied with the information and having all doubts clarified by the physician.
- Giving consent to undergo the surgical procedure and participate in the study, allow the recording of described variables, and analysis of obtained results under proper data protection.

| Signed in Madrid, on the day of20 | Signed in Madrid, on the day of20 |
|-----------------------------------|-----------------------------------|
| Patient or Legal Representative | Physician |

4. Understanding the right to revoke consent at any time without reason and

without affecting medical care.

### **REVOCATION OF CONSENT**

| The | undersigned | patient | hereby | revokes | the | conse | nt given | to | Dr |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | for | the | proposed | sur | gica |
| treatr | ment and inclusi | on in the o | clinical res | earch study | - | | | | |
| This | revocation does | not result | in any pre | ejudice to yo | ur me | dical ca | ıre. | | |
| Signe | ed in Madrid, or | | day of<br>20 | Signe | d in M | adrid, d | on the | _day o<br>20 | of<br> |
| Patie | ent or Legal Rep | resentativ | e | Physi | cian | | | | |

### **CONFIDENTIALITY AND DATA PROTECTION**

All data collected about you and your health during the study will only be used for this purpose. Any future related studies will require prior approval by a Research Ethics Committee.

Your data will be treated with strict confidentiality: your name and personal health information will be replaced with a code. Only the principal investigator will have access to the code. Access to the study data (including health information) will be limited to the research team, study monitor, ethics committee members, and competent health authorities to ensure compliance with laws and regulations.

The data controller is Hospital Clínico San Carlos ("HCSC"), which will take all necessary security measures. Your data will be retained until the end of the study and for 25 years thereafter.

According to Organic Law 3/2018 on the Protection of Personal Data and Digital Rights, you may exercise your rights to access, rectify, oppose, or delete your data. You may also restrict processing of incorrect data, request a copy, or request data portability, if applicable. To exercise these rights, contact the principal investigator (NAME, CENTER, TELEPHONE). You may also contact the Data Protection Agency if dissatisfied. More information: https://www.aepd.es/guias/guia-ciudadano.pdf

### **HCSC Data Protection Officer Contact:**

Secretary of the Data Protection Delegate Committee Calle Melchor Fernández Almagro, 1, 28029 Madrid

Email: protecciondedatos.sanidad@madrid.org

Annex 3. Morphological Classification (Schizas) of Lumbar Spinal Stenosis Based on MRI.



### Annex 4. Zurich Claudication Questionnaire (ZCQ) (Spanish adapted version).

#### Cuestionario de claudicación de Zurich

#### Durante el último mes, ¿cómo describiría...

- ... el dolor que ha experimentado, de media, teniendo en cuenta su dolor de espalda, glúteos y piernas?
  - 1. Ausente
  - 2. Leve
  - 3. Moderado
  - 4. Intenso
  - 5. Muy intenso
- 2) ... cuán a menudo ha experimentado dolor en la espalda, los glúteos o las piernas?
  - 1. Menos de una vez por semana
  - 2. Como mínimo una vez por semana
  - 3. Cada día, durante como mínimo unos minutos
  - 4. Cada día, durante la mayor parte del día
  - 5. Cada día, a todas horas
- 3) ... el dolor que ha sentido en la espalda o los glúteos?
  - 1. Ausente
  - 2. Leve
  - 3. Moderado
  - 4. Intenso
  - 5. Muy intenso
- 4) ... el dolor que ha sentido en las piernas o los pies?
  - 1. Ausente
  - 2. Leve
  - 3. Moderado
  - 4. Intenso
  - 5. Muy intenso
- 5) ... el entumecimiento u hormigueo que ha sentido en las piernas o pies?
  - 1. Ausente
  - 2. Leve
  - 3. Moderado
  - 4. Intenso
  - 5. Muy intenso
- 6) ... la debilidad que ha sentido en las piernas o pies?
  - 1. Ausente
  - 2. Leve
  - 3. Moderada
  - 4. Intensa
  - 5. Muy intensa
- 7) ... sus problemas de equilibrio?
  - 1. No, no he tenido problemas de equilibrio.
    - Sí, a veces me falta el equilibrio o no me siento con paso firme.
    - Sí, a menudo me falta el equilibrio o no me siento con paso firme.

### Durante el último mes, en un día normal...

- 8) ... ¿cuánto ha sido capaz de caminar?
  - 1. Más de 3 km o una hora
  - 2. Más de un par de manzanas, pero menos de 3 km o menos de una hora
  - 3. Más de 15 metros, pero menos de un par de manzanas
  - 4. Menos de 15 metros

- 9) ... ¿ha salido a pasear o ha ido a centros comerciales por placer?
  - 1. Sí, sin problemas
  - 2. Sí, aunque a veces con dolor
  - 3. Sí, pero siempre con dolor
  - 4 No
- 10) ... ¿ha ido a hacer la compra o de tiendas?
  - 1. Sí, sin problemas
  - 2. Sí, aunque a veces con dolor
  - 3. Sí, pero siempre con dolor
  - 4. No
- 11) ... ¿ha caminado por las diferentes habitaciones de su casa o apartamento?
  - 1. Sí, sin problemas
  - 2. Sí, aunque a veces con dolor
  - 3. Sí, pero siempre con dolor
  - 4. No
- 12) ... ¿ha caminado desde su dormitorio hasta el baño?
  - 1. Sí, sin problemas
  - 2. Sí, aunque a veces con dolor
  - 3. Sí, pero siempre con dolor
  - 4. No

#### ¿Cómo está de satisfecho con...

- 13) ... el resultado global de su operación de espalda?
  - 1. Muy satisfecho/a
  - 2. Satisfecho/a
  - 3. Insatisfecho/a
  - 4. Muy insatisfecho/a
- 14) ... el alivio del dolor después de la operación?
  - 1. Muy satisfecho/a
  - 2. Satisfecho/a
  - 3. Insatisfecho/a
  - 4. Muy insatisfecho/a
- 15) ... su capacidad de caminar después de la operación?
  - 1. Muy satisfecho/a
  - 2. Satisfecho/a
  - 3. Insatisfecho/a
  - 4. Muy insatisfecho/a
- 16) ... su capacidad de realizar su trabajo habitual, tareas domésticas o trabajos de jardinería?
  - 1. Muy satisfecho/a
  - 2. Satisfecho/a
  - 3. Insatisfecho/a
  - 4. Muy insatisfecho/a
- 17) ... la fuerza de sus muslos, piernas y pies?
  - 1. Muy satisfecho/a
  - 2. Satisfecho/a
  - 3. Insatisfecho/a
  - 4. Muy insatisfecho/a
- 18) ... su equilibrio o la firmeza de su paso?
  - 1. Muy satisfecho/a
  - 2. Satisfecho/a
  - 3. Insatisfecho/a
  - 4. Muy insatisfecho/a

### Annex 5. Numeric Pain Rating Scale (NPRS).



### Annex 6. Owestry Disability Index (ODI).

| Section | 1 - Pain intensity | Section 6 – Standing | |
|---|---|---|---|
| | I have no pain at the moment | | I can stand as long as I want without |
| | The pain is very mild at the moment | | extra pain |
| | The pain is moderate at the moment | Ö | I can stand as long as I want but it gives |
| | The pain is fairly severe at the moment | - | me extra pain |
| | The pain is very severe at the moment | i i | Pain prevents me from standing for more |
| - H | . B. H. (1) [1] | 1 | than 1 hour |
| 110 | The pain is the worst imaginable at the<br>moment | | Pain prevents me from standing for more |
| | moment | - 1 | than 30 minutes |
| Section | 2 - Personal care (washing, dressing | 6 | Pain prevents me from standing for more |
| etc.) | | 8 | than 10 minutes |
| | I can look after myself normally without causing extra pain | | Pain prevents me from standing at all |
| | I can look after myself normally but it | Section | 7 – Sleeping |
| 0.54 | causes extra pain | | My sleep is never disturbed by pain |
| 0 | It is painful to look after myself and I am | | My sleep is occasionally disturbed by |
| 100 | slow and careful | | pain |
| | | 8 | Because of pain I have less than 6 hours |
| | I need some help but manage most of my | | 일당 그리아 하다 하다 하다 하다 하다 하다 하나 하다 하나 하다 하나 하나 하나 하나 하나 하나 하다 하다 하다 하다 하다 하나 |
| | personal care | 8 | sleep |
| | I need help every day in most aspects of | | Because of pain I have less than 4 hours |
| | self-care | | sleep |
| | I do not get dressed, I wash with | 8 | Because of pain I have less than 2 hours |
| | difficulty and stay in bed | - 2 | sleep |
| Section | 3 – Lifting | | Pain prevents me from sleeping at all |
| | I can lift heavy weights without extra | Section | 8 - Sex life (if applicable)* |
| | pain | | My sex life is normal and causes no |
| | I can lift heavy weights but it gives extra | | extra pain |
| | pain | 8 | My sex life is normal but causes some |
| ū | Pain prevents me from lifting heavy | | extra pain |
| 11 5.44 | weights off the floor, but I can manage if | | My sex life is nearly normal but is very |
| | they are conveniently placed e.g. on a | - | painful |
| | table | Ö | My sex life is severely restricted by pain |
| | Pain prevents me from lifting heavy | | My sex life is nearly absent because of |
| | weights but I can manage light to | | pain |
| | medium weights if they are conveniently | 0 | ************************************** |
| | positioned | | Pain prevents any sex life at all |
| 0 | I can lift very light weights | Section | 9 – Social life |
| | I cannot lift or carry anything at all | | My social life is normal and gives me no |
| | r cannot int or carry anything at an | | extra pain |
| Section | 4 – Walking | | My social life is normal but increases the |
| | Pain does not prevent me walking any | | degree of pain |
| 3900 | distance | | Pain has no significant effect on my |
| | Pain prevents me from walking more | | social life apart from limiting my more |
| | than 2 kilometres | | energetic interests e.g. sport |
| | Pain prevents me from walking more | | Pain has restricted my social life and I do |
| | than 1 kilometre | | not go out as often |
| D | Pain prevents me from walking more | | Pain has restricted by social life to my |
| | than 500 metres | - F | home |
| | I can only walk using a stick or crutches | | I have no social life because of pain |
| | I am in bed most of the time | 107 2007 | Thave no social me occause of pain |
| 55 2037 | Tain in oca most of the time | Section | 10 – Travelling |
| Section | 5 – Sitting | | I can travel anywhere without pain |
| | I can sit in any chair as long as I like | | I can travel anywhere but it gives me |
| | I can only sit in my favourite chair as | | extra pain |
| | long as I like | | Pain is bad but I manage journeys over |
| | Pain prevents me sitting more than one | | two hours |
| | hour | | Pain restricts me to journeys of less than |
| | Pain prevents me from sitting more than | | one hour |
| | 30 minutes | | Pain restricts me to short necessary |
| D | Pain prevents me from sitting more than | | journeys under 30 minutes |
| | 10 minutes | | Pain prevents me from travelling except |
| П | Pain prevents me from sitting at all | | to receive treatment |
| | 1 | | |

### Annex 7. Japanese Orthopedic Association Back Pain Evaluation Questionnaire (JOABPEQ).

With regard to your health condition during the last week, please circle the one item number of the answer for the following questions that best applies. If your condition varies depending on the day or the time, circle the item number of your condition at its worst.

- Q1-1 To alleviate low back pain, you often change your posture.
- 1) Yes 2) No
- Q1-2 Because of the low back pain, you lie down more often than usual.
- 1) Yes 2) No
- Q1-3 Your lower back is almost always aching.
- 1) Yes 2) No
- Q1-4 Because of the low back pain, you cannot sleep well. (If you take sleeping pills because of the pain, select "No.")
- 1) No 2) Yes
- Q2-1 Because of the low back pain, you sometimes ask someone to help you when you do something.
- 1) Yes 2) No
- Q2-2 Because of the low back pain, you refrain from bending forward or kneeling down.
- 1) Yes 2) No
- Q2-3 Because of the low back pain, you have difficulty in standing up from a chair.
- 1) Yes 2) No
- Q2-4 Because of the low back pain, turning over in bed is difficult.
- 1) Yes 2) No
- Q2-5 Because of the low back pain, you have difficulty putting on socks or stockings.
- 1) Yes 2) No

- Q2-6 Do you have difficulty in any one of the following motions; vending forward, kneeling or stooping?
- 1) I have great difficulty 3) I have no difficulty
- 2) I have some difficulty
- Q3-1 Because of the low back pain, you walk only short distances.
- 1) Yes 2) No
- Q3-2 Because of the low back pain, you stay seated most of the day.
- 1) Yes 2) No
- Q3-3 Because of the low back pain, you go up the stairs more slowly than usual.
- 1) Yes 2) No
- Q3-4 Do you have difficulty in going up the stairs?
- 1) I have great difficulty 2) I have some difficulty 3) I have no difficulty Q3-5 Do you have difficulty in walking more than 15 minutes?
- 1) I have great difficulty 2) I have some difficulty 3) I have no difficulty

# Q4-1 Because of the low back pain, you do not do any routine housework these days.

1) No 2) Yes

# Q4-2 Have you been unable to do your work or ordinary activities as well as you would like?

- 1) I have not been able to do them at all.
- 2) I have been unable to do them most of the time.
- 3) I have sometimes been unable to do them.
- 4) I have been able to do them most of the time.
- 5) I have always been able to do them.

### Q4-3 Has your work routine been hindered because of the pain?

- 1) Greatly 2) Moderately 3) Slightly (somewhat)
- 4) Little (minimally) 5) Not at all

# Q5-1 Because of the low back pain, you get irritated or get angry at other persons more often than usual.

1) Yes 2) No

### Q5-2 How is your present health condition?

- 1) Poor 2) Fair 3) Good 4) Very good
- 5) Excellent

### Q5-3 Have you been discouraged and depressed?

1) Always 2) Frequently 3) Sometimes 4) Rarely 5) Never **Q5-4 Do you feel exhausted?** 

1) Always 2) Frequently 3) Sometimes 4) Rarely 5) Never

### Q5-5 Have you felt happy?

1) Never 2) Rarely 3) Sometimes 4) Almost always 5) Always

### Q5-6 Do you think you are in decent health?

- 1) Not at all (my health is very poor)
- 2) Barely (my health is poor)
- 3) Not very much (my health is average health)
- 4) Fairly (my health is better than average)
- 5) Yes (I am healthy)

### Q5-7 Do you feel your health will get worse?

- 1) Very much so 2) A little bit at a time
- 3) Sometimes yes and sometimes no
- 4) Not very much 5) Not at all

### **Measurement:**

- Social life function: ('Q1-2' × 2 + 'Q2-4' × 4 + 'Q2-5' × 6 + 'Q2-6' × 10 22)
   × 100 ÷ 74
- Mental health: ('Q1-13' × 3 + 'Q2-1' × 4 + 'Q2-7' × 6 + 'Q2-8' × 6 + 'Q2-9' × 3 + 'Q2-10' × 3 + 'Q2-11' × 3 28) × 100 ÷ 103
- Lumbar function:  $('Q1-4' \times 10 + 'Q1-5' \times 10 + 'Q1-6' \times 20 + 'Q1-8' \times 10 + 'Q1-9' \times 30 + 'Q2-3' \times 20 100) \times 100 \div 120$
- Walking ability: ('Q1-10' × 30 + 'Q1-12' × 20 + 'Q1-14' × 10 + 'Q2-2' × 10 + 'Q2-4' × 30 100) × 100 ÷ 140
- Low back pain: ('Q1-1' × 20 + 'Q1-3' × 20 + 'Q1-7' × 20 + 'Q1-11' × 10 70) × 100 ÷ 70